CLINICAL TRIAL: NCT01807923
Title: A Phase 3, Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Lumacaftor in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Homozygous for the F508del CFTR Mutation
Brief Title: A Study of Lumacaftor in Combination With Ivacaftor in Cystic Fibrosis Subjects Aged 12 Years and Older Who Are Homozygous for the F508del-CFTR Mutation
Acronym: TRAFFIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX12-809-103
Record Dates: First submitted 2013-03-04; First posted 2013-03-08 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-06

CONDITIONS: Cystic Fibrosis, Homozygous for the F508del CFTR Mutation
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo matched to lumacaftor (LUM, VX-809) and ivacaftor (IVA, VX-770) tablet every 12 hours (q12h), up to Week 24.
  Interventions: Drug: Placebo
- LUM 600 mg qd/IVA 250 mg q12h (Experimental): LUM 600 milligram (mg) plus IVA 250 mg fixed-dose combination (FDC) tablet in the morning and IVA 250 mg film-coated tablet in the evening, up to Week 24.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination; Drug: Ivacaftor
- LUM 400 mg q12h/ IVA 250 mg q12h (Experimental): LUM 400 mg plus IVA 250 mg FDC tablet in the morning and in the evening, up to Week 24.
  Interventions: Drug: Lumacaftor Plus Ivacaftor Combination

INTERVENTIONS:
Drug: Lumacaftor Plus Ivacaftor Combination — Fixed dose combination tablet
  Other Names: VX-809+VX-770, LUM+IVA
  Arms: LUM 400 mg q12h/ IVA 250 mg q12h; LUM 600 mg qd/IVA 250 mg q12h
Drug: Ivacaftor — Film-coated tablet
  Other Names: VX-770, IVA
  Arms: LUM 600 mg qd/IVA 250 mg q12h
Drug: Placebo — Matching placebo tablet
  Arms: Placebo

SUMMARY:
The primary objective of the study was to evaluate the efficacy of lumacaftor in combination with ivacaftor at Week 24 in participants aged 12 years and older with cystic fibrosis (CF) who are homozygous for the F508del mutation on the CF transmembrane conductance regulator (CFTR) gene.

DETAILED DESCRIPTION:
This was a Phase 3, randomized, double-blind, placebo-controlled, parallel-group multicenter study of orally administered lumacaftor in combination with ivacaftor in participants aged 12 years and older with CF who are homozygous for the F508del-CFTR mutation.

The study included a Screening Period (Day -28 through Day -1), a Treatment Period (Day 1 [first dose of study drug] to Week 24 ± 5 days), and a Safety Follow-up Visit (4 weeks ± 7 days after the Week 24 Visit).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Homozygous for the F508del CFTR mutation
* Forced expiratory volume in 1 second (FEV1) greater than or equal to (>=) 40 percent (%) and less than or equal to (=<) 90% of predicted normal for age, sex, and height
* Willing to remain on a stable CF medication regimen through Week 24 or, if applicable, the Safety Follow up Visit

Exclusion Criteria:

* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 4 weeks before first dose of study drug
* History of solid organ or hematological transplantation
* History of alcohol or drug abuse in the past year
* Ongoing or prior participation in an investigational drug study (including studies investigating lumacaftor and/or ivacaftor) within 30 days of screening
* Use of strong inhibitors, moderate inducers or strong inducers of Cytochrome P450 3A (CYP3A) within 14 days before Day 1 of dosing

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (89):
- United States (48):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Fresno, California
  - La Jolla, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Madera, California
  - Oakland, California
  - Palo Alto, California
  - Denver, Colorado
  - Gainsville, Florida
  - Hollywood, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Peoria, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Kansas City, Missouri
  - Bedford, New Hampshire
  - Lebanon, New Hampshire
  - Long Branch, New Jersey
  - Hawthorne, New York
  - New York, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Knoxville, Tennessee
  - Austin, Texas
  - Tyler, Texas
  - Colchester, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
- Australia (3):
  - Broadmeadow, New South Wales
  - Westmead, New South Wales
  - Adelaide, South Australia
- Canada (4):
  - Halifax, British Columbia
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
- Czechia (3):
  - Brno
  - Plzen-Bory
  - Prague
- France (5):
  - Strasbourg, Bas Rhin
  - Roscoff, Finistere
  - Paris, Paris
  - Bron, Rhone
  - Pierre-Bénite, Rhone
- Germany (6):
  - Tübingen, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Würzburg, Bavaria
  - Cologne, North Rhine-Westphalia
  - Leipzig, Saxony
  - Berlin, State of Berlin
- Ireland (2):
  - Dublin, Dublin
  - Tallaght, Dublin
- Italy (6):
  - Florence, Firenze
  - Ancona
  - Genova
  - Milan
  - Roma
  - Verona
- Netherlands (4):
  - Amsterdam
  - Nijmegen
  - Rotterdam
  - The Hague
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala
- United Kingdom (5):
  - Belfast, Belfast
  - Exeter, Devon
  - Southhampton, Hampshire
  - Nottingham, Nottinghamshire
  - Birmingham, West Midlands

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Acaster S, Mukuria C, Rowen D, Brazier JE, Wainwright CE, Quon BS, Duckers J, Quittner AL, Lou Y, Sosnay PR, McGarry LJ. Development of the Cystic Fibrosis Questionnaire-Revised-8 Dimensions: Estimating Utilities From the Cystic Fibrosis Questionnaire-Revised. Value Health. 2023 Apr;26(4):567-578. doi: 10.1016/j.jval.2022.12.002. Epub 2022 Dec 9. PMID 36509366
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Flume PA, Suthoff ED, Kosinski M, Marigowda G, Quittner AL. Measuring recovery in health-related quality of life during and after pulmonary exacerbations in patients with cystic fibrosis. J Cyst Fibros. 2019 Sep;18(5):737-742. doi: 10.1016/j.jcf.2018.12.004. Epub 2018 Dec 23. PMID 30587335
- [Derived] McColley SA, Konstan MW, Ramsey BW, Stuart Elborn J, Boyle MP, Wainwright CE, Waltz D, Vera-Llonch M, Marigowda G, Jiang JG, Rubin JL. Lumacaftor/Ivacaftor reduces pulmonary exacerbations in patients irrespective of initial changes in FEV1. J Cyst Fibros. 2019 Jan;18(1):94-101. doi: 10.1016/j.jcf.2018.07.011. Epub 2018 Aug 23. PMID 30146268
- [Derived] Elborn JS, Ramsey BW, Boyle MP, Konstan MW, Huang X, Marigowda G, Waltz D, Wainwright CE; VX-809 TRAFFIC and TRANSPORT study groups. Efficacy and safety of lumacaftor/ivacaftor combination therapy in patients with cystic fibrosis homozygous for Phe508del CFTR by pulmonary function subgroup: a pooled analysis. Lancet Respir Med. 2016 Aug;4(8):617-626. doi: 10.1016/S2213-2600(16)30121-7. Epub 2016 Jun 10. PMID 27298017
- [Derived] Wainwright CE, Elborn JS, Ramsey BW, Marigowda G, Huang X, Cipolli M, Colombo C, Davies JC, De Boeck K, Flume PA, Konstan MW, McColley SA, McCoy K, McKone EF, Munck A, Ratjen F, Rowe SM, Waltz D, Boyle MP; TRAFFIC Study Group; TRANSPORT Study Group. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Jul 16;373(3):220-31. doi: 10.1056/NEJMoa1409547. Epub 2015 May 17. PMID 25981758

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Started | 187 | 185 | 187
Completed | 182 | 179 | 176
Not Completed | 5 | 6 | 11
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Withdrawal of Consent (not due to AE) | 0 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Not Eligible (Genotype) | 0 | 0 | 1
Not completed — Randomized But Not Treated | 3 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received any amount of study drug.
Groups:
- Placebo: Placebo matched to LUM and IVA tablet q12h, up to Week 24.
- LUM 600 mg qd/IVA 250 mg q12h: LUM 600 mg plus IVA 250 mg FDC tablet in the morning and IVA 250 mg film-coated tablet in the evening, up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h | Total
Number analyzed (Participants) | 184 | 183 | 182 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (10.80) | 24.7 (9.71) | 25.5 (10.09) | 25.1 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 86 | 84 | 254
  Male | 100 | 97 | 98 | 295

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at Week 24
Description: Absolute change from baseline at Week 24 was assessed as the average treatment effect at Week 16 and at Week 24. FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, race, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years.
Time Frame: Baseline, Week 16 and 24
Population: Full Analysis Set (FAS) included all randomized participants who received any amount of study drug. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 180 | 176 | 172
percent predicted of FEV1 | -0.44 (0.524) | 3.59 (0.525) | 2.16 (0.530)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using mixed-effects model for repeated measures (MMRM) model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (less than (<)18 versus greater than equal to (>=18) years old), and percent predicted FEV1 severity at Screening (<70 versus >=70); Test type: Superiority or Other; p < 0.0001, MMRM; Least Squares (LS) Mean Difference = 4.03, 95% CI 2-sided [2.62 to 5.44]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed using MMRM model, as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0003, MMRM; LS Mean Difference = 2.60, 95% CI 2-sided [1.18 to 4.01]

2. Secondary Outcome: Relative Change From Baseline in Percent Predicted FEV1 at Week 24
Description: Assessed as the average treatment effect at Week 16 and at Week 24. FEV1 and percent predicted FEV1 are defined in Outcome Measure (OM) 1.
Time Frame: Baseline, Week 16 and 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 180 | 176 | 172
percent change | -0.34 (0.913) | 6.39 (0.914) | 3.99 (0.923)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), and percent predicted FEV1 severity at Screening (<70 versus >=70); Test type: Superiority or Other; p < 0.0001, MMRM; LS Mean Difference = 6.73, 95% CI 2-sided [4.27 to 9.19]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed using MMRM model, as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0006, MMRM; LS Mean Difference = 4.33, 95% CI 2-sided [1.86 to 6.80]

3. Secondary Outcome: Absolute Change From Baseline in Body Mass Index (BMI) at Week 24
Description: BMI was defined as weight in kilogram (kg) divided by height*height in square meter (m^2).
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kilogram per square meter (kg/m^2)
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 178 | 176
kilogram per square meter (kg/m^2) | 0.19 (0.070) | 0.35 (0.070) | 0.32 (0.071)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline BMI; Test type: Superiority or Other; p = 0.1122, MMRM; LS Mean Difference = 0.16, 95% CI 2-sided [-0.04 to 0.35]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed using MMRM model, as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.1938, MMRM; LS Mean Difference = 0.13, 95% CI 2-sided [-0.07 to 0.32]

4. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score at Week 24
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), the scaled score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 176 | 172
units on a scale | 1.10 (1.161) | 4.98 (1.178) | 2.60 (1.192)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline CFQ-R respiratory domain score; Test type: Superiority or Other; p = 0.0168, MMRM — This test is considered nominally significant because a hierarchical procedure was used and was broken prior to this test; LS Mean Difference = 3.88, 95% CI 2-sided [0.70 to 7.05]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed using MMRM model, as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.3569, MMRM; LS Mean Difference = 1.50, 95% CI 2-sided [-1.69 to 4.69]

5. Secondary Outcome: Percentage of Participants With Response Based on Percent Predicted FEV1
Description: A participant was considered as a responder if the participant had >=5% increase from baseline in average percent predicted FEV1 at Week 16 and at Week 24 (relative change). FEV1 and percent predicted FEV1 are defined in OM 1. A participant with a missing average relative change from baseline in percent predicted FEV1 at Week 16 and at Week 24 was considered as a non-responder.
Time Frame: Week 16 and 24
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 183 | 182
percentage of participants | 22.3 | 46.4 | 36.8
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Odds Ratio (OR) and 95% confidence intervals (Cis) are Mantel-Haenszel estimates. P values are from a Cochran-Mantel-Haenszel test stratified by sex (male versus female), age group at baseline (<18 versus >=18 years old), and percent predicted FEV1 severity at Screening (<70 versus >=70); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.9378, 95% CI 2-sided [1.8786 to 4.5941]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0023, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.0592, 95% CI 2-sided [1.2920 to 3.2819]

6. Secondary Outcome: Number of Pulmonary Exacerbation Events
Description: The total number of days on study is equal to the Week 24 date or the last dose date (whichever occurred last) minus the first dose date plus 1. The total number of years (48 weeks) on study is equal to the number of days on study divided by 336. Pulmonary exacerbation events per year (48 weeks) are reported.
Time Frame: through Week 24
Population: FAS.
Measure: Number; unit: pulmonary exacerbation events per year
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 183 | 182
pulmonary exacerbation events per year | 1.07 | 0.77 | 0.71
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using regression analysis for a negative binomial distribution with sex (male versus female), age group at baseline (<18 versus >=18 years old), and percent predicted FEV1 severity at Screening (<70 versus >=70) as covariates with the logarithm of time on study as the offset; Test type: Superiority or Other; p = 0.0491, Negative Binomial Regression; Event Rate Ratio = 0.7186, 95% CI 2-sided [0.5170 to 0.9987]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0169, Negative Binomial Regression — [p-value comment as in outcome 4, analysis 1]; Event Rate Ratio = 0.6643, 95% CI 2-sided [0.4749 to 0.9291]

7. Secondary Outcome: Absolute Change From Baseline in Weight at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 178 | 176
kilograms (kg) | 0.93 (0.202) | 1.34 (0.205) | 1.23 (0.205)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline weight; Test type: Superiority or Other; p = 0.1565, MMRM; LS Mean Difference = 0.40, 95% CI 2-sided [-0.16 to 0.96]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.2992, MMRM; LS Mean Difference = 0.30, 95% CI 2-sided [-0.26 to 0.86]

8. Secondary Outcome: Absolute Change From Baseline in BMI-for-age Z-score at Week 24
Description: Z-Score is a statistical measure to evaluate how a single data point compares to a standard. It describes whether a mean was above or below the standard and how unusual the measurement is with range from -infinity to + infinity; 0: same mean, >0: a greater mean, and <0: a lesser mean than the standard. BMI-for-age z-score was calculated by using Centers for Disease Control and Prevention (CDC) growth charts for the pediatric population.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Only participants who were <20 years of age were analyzed.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 69 | 65 | 58
z-score | 0.0153 (0.04886) | 0.1132 (0.05081) | 0.0933 (0.05431)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline BMI z-score; Test type: Superiority or Other; p = 0.1539, MMRM; LS Mean Difference = 0.0980, 95% CI 2-sided [-0.0370 to 0.2330]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.2713, MMRM; LS Mean Difference = 0.0781, 95% CI 2-sided [-0.0615 to 0.2176]

9. Secondary Outcome: Time-to-First Pulmonary Exacerbation
Description: Time to first pulmonary exacerbation was assessed using Cox Regression. For participants who completed 24 weeks of treatment, participants without a pulmonary exacerbation before treatment completion were considered censored at the time of treatment completion or at the Week 24 Visit (whichever occurred last). For participants who prematurely discontinued study treatment, participants without a pulmonary exacerbation through the Week 24 Visit were considered censored at the time of the Week 24 Visit.
Time Frame: through Week 24
Population: FAS.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 183 | 182
days | NA [NA to NA] — Median time was not reached as less than 50% of participants had the event of interest. | NA [NA to NA] — Median time was not reached as less than 50% of participants had the event of interest. | NA [NA to NA] — Median time was not reached as less than 50% of participants had the event of interest.
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using Cox proportional hazard regression, time is the time-to-first event or censoring, with adjustment for sex (male versus female), age group at baseline (<18 versus >=18 years old), and percent predicted FEV1 severity at Screening (<70 versus >=70); Test type: Superiority or Other; p = 0.0396, Cox Proportional Hazard Regression; Hazard Ratio (HR) = 0.692
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0385, Cox Proportional Hazard Regression; Hazard Ratio (HR) = 0.691

10. Secondary Outcome: Percentage of Participants With At Least 1 Pulmonary Exacerbation Event
Time Frame: through Week 24
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 183 | 182
percentage of participants | 39.7 | 30.1 | 30.2
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; OR and 95% confidence intervals (CIs) are Mantel-Haenszel estimates. P values are from a Cochran-Mantel-Haenszel test stratified by sex (male versus female), age group at baseline (<18 versus >=18 years old), and percent predicted FEV1 severity at Screening (<70 versus >=70); Test type: Superiority or Other; p = 0.0552, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.6565, 95% CI 2-sided [0.4266 to 1.0103]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0512, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.6438, 95% CI 2-sided [0.4142 to 1.0005]

11. Secondary Outcome: Absolute Change From Baseline in Euro Quality of Life Scale (EuroQol) 5-Dimension-3 Level (EQ-5D-3L) Index Score at Week 24
Description: EQ-5D-3L: participant rated questionnaire to assess health-related quality of life. It consists of EQ-5D descriptive system and EQ-5D Visual Analog Scale (VAS). EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). The 5 dimensional 3-level systems are converted into a single index utility score. Values for theoretically possible health states are calculated using a regression model and weighted according to the social preferences of the Unites States (US) general population. For this population, the possible EQ-5D-3L index scores ranges from -0.11 (that is, 3 for all 5 dimensions) to 1.0 (that is, 1 for all 5 dimensions), where higher scores indicate a better health state.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 179 | 175 | 170
units on a scale | 0.0006 (0.00739) | 0.0066 (0.00746) | 0.0100 (0.00757)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline EQ-5D-3L index score; Test type: Superiority or Other; p = 0.5604, MMRM; LS Mean Difference = 0.0060, 95% CI 2-sided [-0.0142 to 0.0262]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.3613, MMRM; LS Mean Difference = 0.0095, 95% CI 2-sided [-0.0109 to 0.0298]

12. Secondary Outcome: Absolute Change From Baseline in EQ-5D-3L VAS Score at Week 24
Description: The EQ-5D-3L VAS records the participant's self-rated health on a vertical, visual analogue scale where the best state a participant can imagine is marked 100 and the worst state a participant can imagine is marked 0, higher scores indicates a better health state.
Time Frame: Baseline, Week 24
Population: FAS. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 180 | 173 | 171
units on a scale | 1.4 (1.03) | 3.5 (1.04) | 2.8 (1.04)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline EQ-5D-3L VAS score; Test type: Superiority or Other; p = 0.1342, MMRM; LS Mean Difference = 2.1, 95% CI 2-sided [-0.7 to 4.9]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.3071, MMRM; LS Mean Difference = 1.4, 95% CI 2-sided [-1.3 to 4.2]

13. Secondary Outcome: Absolute Change From Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Domain Scores at Week 24
Description: The TSQM is a 14-item self-administered questionnaire which measures participants' experiences with their medication on four dimensions: effectiveness, side effects, convenience and global satisfaction. For each dimension, responses are added and transformed to a scale from 0 to 100, where higher scores indicate greater satisfaction.
Time Frame: Baseline, Week 24
Population: FAS. Here, "n" signifies participants who were evaluable for specified category for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 183 | 182
units on a scale
  Effectiveness (n = 163, 156, 144) | -5.30 (1.643) | 0.19 (1.666) | 0.50 (1.726)
  Side Effects (n = 162, 154, 143) | 2.23 (1.119) | -1.94 (1.141) | -2.51 (1.179)
  Convenience (n = 163, 154, 144) | 4.37 (1.504) | 4.98 (1.540) | 7.45 (1.579)
  Global Satisfaction (n= 163, 154, 144) | -10.49 (1.863) | -5.00 (1.906) | -3.77 (1.956)
Statistical Analysis 1: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Effectiveness: analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline TSQM effectiveness score; Test type: Superiority or Other; p = 0.0160, MMRM; LS Mean Difference = 5.49, 95% CI 2-sided [1.03 to 9.96]
Statistical Analysis 2: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Effectiveness: analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0126, MMRM; LS Mean Difference = 5.80, 95% CI 2-sided [1.25 to 10.35]
Statistical Analysis 3: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Side Effects: analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline TSQM side effects score; Test type: Superiority or Other; p = 0.0074, MMRM; LS Mean Difference = -4.18, 95% CI 2-sided [-7.23 to -1.13]
Statistical Analysis 4: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Side Effects: analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0029, MMRM; LS Mean Difference = -4.74, 95% CI 2-sided [-7.85 to -1.63]
Statistical Analysis 5: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Convenience: analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline TSQM convenience score; Test type: Superiority or Other; p = 0.7721, MMRM; LS Mean Difference = 0.61, 95% CI 2-sided [-3.50 to 4.71]
Statistical Analysis 6: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Convenience: analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.1472, MMRM; LS Mean Difference = 3.08, 95% CI 2-sided [-1.09 to 7.25]
Statistical Analysis 7: Comparison: Placebo vs LUM 600 mg qd/IVA 250 mg q12h; Global Satisfaction: analysis was performed using MMRM model including treatment, visit, and treatment-by-visit interaction as fixed effects with adjustments for sex (male versus female), age group at baseline (<18 versus >=18 years old), percent predicted FEV1 severity at Screening (<70 versus >=70), and baseline TSQM global satisfaction score; Test type: Superiority or Other; p = 0.0345, MMRM; LS Mean Difference = 5.49, 95% CI 2-sided [0.40 to 10.58]
Statistical Analysis 8: Comparison: Placebo vs LUM 400 mg q12h/ IVA 250 mg q12h; Global Satisfaction: analysis was performed as described in Statistical Analysis 1; Test type: Superiority or Other; p = 0.0109, MMRM; LS Mean Difference = 6.72, 95% CI 2-sided [1.55 to 11.89]

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Treatment-Emergent Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes serious as well as Nonserious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Any AE that increased in severity or that was newly developed at or after the initial dosing of study drug to 28 days after the last dose of study drug is considered treatment-emergent.
Time Frame: up to Week 28
Population: Safety Set (SS) included all randomized participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 184 | 183 | 182
participants
  Participants With Treatment-Emergent AEs | 174 | 175 | 174
  Participants With Treatment-Emergent SAEs | 49 | 33 | 33

15. Secondary Outcome: Pre-dose Concentration (Ctrough), Average Pre-dose Concentration (Ctrough,Avg), 3 to 6 Hours Post-dose Concentration (C3-6h), and Average 3 to 6 Hours Post-dose Concentration (C3-6h,Avg)
Description: Ctrough, Ctrough, avg, C3-6h, and C3-6h, avg for lumacaftor, M28 lumacaftor (lumacaftor metabolite), ivacaftor, M1 ivacaftor (ivacaftor metabolite), and M6 ivacaftor (ivacaftor metabolite) were calculated. C3-6h,ave is average of individual 3 to 6 hours post-dose observed concentrations across Day 15, and Weeks 4 and 8 and Ctrough, ave is average of individual pre-dose observed concentrations across Weeks 4, 8, and 16. This outcome was not planned to be assessed in Placebo arm.
Time Frame: For C3-6h: 3 to 6 hours after morning dose on Day 1 and 15, Week 4 and 8; For C3-6h,avg 3 to 6 hours after morning dose on Day 15, Week 4 and 8; For Ctrough and Ctrough,avg: before morning dose on Week 4, 8, and 16
Population: Pharmacokinetic (PK) population included all randomized participants who received at least one dose of study drug and had a PK assessment. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure and "n" signifies participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Number analyzed (Participants) | 180 | 181
microgram per milliliter (mcg/mL)
  LUM, Day 1: C3-6h (n = 180, 175) | 27.5 (12.5) | 18.4 (8.55)
  LUM, Day 15: Ctrough (n = 172, 175) | 7.56 (5.33) | 14.1 (6.99)
  LUM, Day 15: C3-6 (n = 167, 171) | 26.1 (11.5) | 23.6 (8.54)
  LUM, Week 4: Ctrough (n = 172, 178) | 7.75 (5.05) | 13.4 (6.70)
  LUM, Week 4: C3-6 (n = 170, 171) | 28.4 (11.2) | 24.2 (8.66)
  LUM, Week 8: Ctrough (n = 173, 174) | 7.43 (5.60) | 13.4 (6.68)
  LUM, Week 8: C3-6 (n = 165, 171) | 28.2 (11.2) | 24.4 (8.80)
  LUM, Week 16: Ctrough (n = 165, 164) | 6.95 (4.99) | 13.5 (7.49)
  M-28 LUM, Day 1: C3-6h (n = 180, 175) | 0.220 (0.107) | 0.179 (0.0811)
  M-28 LUM, Day 15: Ctrough (n = 172, 175) | 1.25 (0.614) | 1.48 (0.590)
  M-28 LUM, Day 15: C3-6 (n = 167, 171) | 1.37 (0.606) | 1.49 (0.576)
  M-28 LUM, Week 4: Ctrough (n = 172, 178) | 1.31 (0.646) | 1.48 (0.642)
  M-28 LUM, Week 4: C3-6 (n = 170, 171) | 1.39 (0.635) | 1.49 (0.615)
  M-28 LUM, Week 8: Ctrough (n = 173, 174) | 1.32 (0.684) | 1.53 (0.674)
  M-28 LUM, Week 8: C3-6 (n = 165, 171) | 1.42 (0.658) | 1.56 (0.669)
  M-28 LUM, Week 16: Ctrough (n = 165, 164) | 1.30 (0.769) | 1.57 (0.757)
  IVA, Day 1: C3-6h (n = 180, 175) | 1.29 (0.624) | 1.24 (0.630)
  IVA, Day 15: Ctrough (n = 172, 176) | 0.151 (0.123) | 0.115 (0.123)
  IVA, Day 15: C3-6 (n = 167, 171) | 0.557 (0.311) | 0.413 (0.199)
  IVA, Week 4: Ctrough (n = 172, 178) | 0.142 (0.107) | 0.105 (0.083)
  IVA, Week 4: C3-6 (n = 170, 171) | 0.638 (0.325) | 0.456 (0.235)
  IVA, Week 8: Ctrough (n = 173, 174) | 0.130 (0.101) | 0.0894 (0.0726)
  IVA, Week 8: C3-6 (n = 165, 171) | 0.648 (0.364) | 0.470 (0.295)
  IVA, Week 16: Ctrough (n = 165, 164) | 0.133 (0.131) | 0.0834 (0.0622)
  M-1 IVA, Day 1: C3-6h (n = 180, 175) | 2.46 (1.29) | 2.41 (1.35)
  M-1 IVA, Day 15: Ctrough (n = 172, 176) | 0.665 (0.578) | 0.511 (0.530)
  M-1 IVA, Day 15: C3-6 (n = 167, 171) | 1.94 (0.981) | 1.71 (0.867)
  M-1 IVA, Week 4: Ctrough (n = 172, 178) | 0.628 (0.492) | 0.450 (0.345)
  M-1 IVA, Week 4: C3-6 (n = 170, 171) | 2.21 (1.01) | 1.76 (0.932)
  M-1 IVA, Week 8: Ctrough (n = 173, 174) | 0.584 (0.451) | 0.404 (0.381)
  M-1 IVA, Week 8: C3-6 (n = 165, 171) | 2.17 (1.06) | 1.78 (0.975)
  M-1 IVA, Week 16: Ctrough (n = 165, 164) | 0.589 (0.519) | 0.396 (0.319)
  M-6 IVA, Day 1: C3-6h (n = 180, 175) | 0.976 (0.877) | 0.927 (0.875)
  M-6 IVA, Day 15: Ctrough (n = 172, 176) | 1.68 (1.31) | 1.67 (1.40)
  M-6 IVA, Day 15: C3-6 (n = 167, 171) | 3.03 (1.96) | 2.87 (1.81)
  M-6 IVA, Week 4: Ctrough (n = 172, 178) | 1.66 (1.36) | 1.46 (0.938)
  M-6 IVA, Week 4: C3-6 (n = 170, 171) | 3.07 (1.92) | 2.49 (1.53)
  M-6 IVA, Week 8: Ctrough (n = 173, 174) | 1.52 (1.12) | 1.31 (0.946)
  M-6 IVA, Week 8: C3-6 (n = 165, 171) | 2.96 (1.86) | 2.36 (1.57)
  M-6 IVA, Week 16: Ctrough (n = 165, 164) | 1.40 (1.11) | 1.33 (1.02)
  LUM: Ctrough,ave (n = 179, 181) | 7.49 (3.93) | 13.5 (5.52)
  LUM: C3-6h,ave (n = 179, 181) | 27.7 (8.63) | 24.0 (7.29)
  M-28 LUM: Ctrough,ave (n = 179, 181) | 1.31 (0.628) | 1.51 (0.614)
  M-28 LUM: C3-6h,ave (n = 179, 181) | 1.39 (0.596) | 1.51 (0.585)
  IVA: Ctrough,ave (n = 179, 181) | 0.137 (0.0773) | 0.0989 (0.0644)
  IVA: C3-6h,ave (n = 179, 181) | 0.614 (0.271) | 0.445 (0.193)
  M1-IVA: Ctrough,ave (n = 179, 181) | 0.606 (0.350) | 0.441 (0.293)
  M1-IVA: C3-6h,ave (n = 179, 181) | 2.11 (0.817) | 1.74 (0.726)
  M6-IVA: Ctrough,ave (n = 179, 181) | 1.57 (0.992) | 1.44 (0.861)
  M6-IVA: C3-6h,ave (n = 179, 181) | 3.04 (1.55) | 2.57 (1.34)

ADVERSE EVENTS:
Time Frame: Up to Week 28
Description: Participants were analyzed as per actual treatment received. Other adverse events includes only non-serious AEs.
Arm/Group | Placebo | LUM 600 mg qd/IVA 250 mg q12h | LUM 400 mg q12h/ IVA 250 mg q12h
Serious Adverse Events (participants affected / at risk) | 49/184 | 33/183 | 33/182
Other Adverse Events (participants affected / at risk) | 173/184 | 175/183 | 172/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | LUM 600 mg qd/IVA 250 mg q12h (N=183) | LUM 400 mg q12h/ IVA 250 mg q12h (N=182)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 41 | 19 | 17
Influenza (Infections and infestations) | 1 | 2 | 0
Tracheobronchitis (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Forced expiratory volume decreased (Investigations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Implant site thrombosis (General disorders) | 0 | 2 | 0
Device dislocation (General disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | LUM 600 mg qd/IVA 250 mg q12h (N=183) | LUM 400 mg q12h/ IVA 250 mg q12h (N=182)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 58 | 57 | 54
Nasopharyngitis (Infections and infestations) | 20 | 9 | 26
Upper respiratory tract infection (Infections and infestations) | 10 | 16 | 17
Viral upper respiratory tract infection (Infections and infestations) | 12 | 15 | 13
Rhinitis (Infections and infestations) | 12 | 16 | 8
Sinusitis (Infections and infestations) | 12 | 7 | 5
Influenza (Infections and infestations) | 3 | 8 | 8
Bronchitis (Infections and infestations) | 7 | 9 | 2
Respiratory tract infection (Infections and infestations) | 3 | 2 | 6
Pharyngitis (Infections and infestations) | 2 | 4 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 4 | 2 | 3
Oral candidiasis (Infections and infestations) | 3 | 2 | 3
Urinary tract infection (Infections and infestations) | 3 | 2 | 3
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 2 | 3
Viral infection (Infections and infestations) | 4 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 2 | 2
Lower respiratory tract infection bacterial (Infections and infestations) | 3 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 3
H1N1 influenza (Infections and infestations) | 1 | 1 | 2
Oral herpes (Infections and infestations) | 1 | 1 | 2
Otitis media (Infections and infestations) | 0 | 3 | 1
Acute sinusitis (Infections and infestations) | 1 | 1 | 1
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 | 2 | 0
Fungal skin infection (Infections and infestations) | 2 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 2 | 0
Sputum purulent (Infections and infestations) | 0 | 2 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 1 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 2 | 0
Mycobacterium abscessus infection (Infections and infestations) | 2 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1
Genital infection fungal (Infections and infestations) | 0 | 1 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 1
Herpes dermatitis (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Overgrowth bacterial (Infections and infestations) | 1 | 0 | 0
Pseudomonas bronchitis (Infections and infestations) | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0
Viral rhinitis (Infections and infestations) | 0 | 1 | 0
Viral tonsillitis (Infections and infestations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 52 | 47
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 23 | 22 | 26
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 23 | 15 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 21 | 17
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 9 | 26 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 25 | 9 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 24 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 5
Rales (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 7
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal exudate (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 16 | 24
Abdominal pain (Gastrointestinal disorders) | 12 | 11 | 23
Nausea (Gastrointestinal disorders) | 11 | 9 | 14
Constipation (Gastrointestinal disorders) | 11 | 6 | 7
Abdominal pain upper (Gastrointestinal disorders) | 10 | 7 | 5
Flatulence (Gastrointestinal disorders) | 1 | 9 | 11
Vomiting (Gastrointestinal disorders) | 2 | 8 | 7
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3 | 3
Enteritis (Gastrointestinal disorders) | 2 | 0 | 3
Steatorrhoea (Gastrointestinal disorders) | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 2 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0
Colonic haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0
Gingivitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 10 | 10 | 13
Bacterial test positive (Investigations) | 9 | 4 | 7
Alanine aminotransferase increased (Investigations) | 5 | 4 | 3
Forced expiratory volume decreased (Investigations) | 7 | 3 | 1
Weight decreased (Investigations) | 5 | 2 | 4
Liver function test abnormal (Investigations) | 6 | 3 | 1
Pulmonary function test decreased (Investigations) | 6 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 3
Blood creatinine increased (Investigations) | 4 | 3 | 1
White blood cell count increased (Investigations) | 1 | 2 | 2
Blood glucose decreased (Investigations) | 3 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 2 | 2
Vitamin D decreased (Investigations) | 1 | 1 | 2
Breath sounds abnormal (Investigations) | 1 | 2 | 0
Fungal test positive (Investigations) | 1 | 1 | 1
Staphylococcus test positive (Investigations) | 0 | 1 | 2
Transaminases increased (Investigations) | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0
Blood immunoglobulin E increased (Investigations) | 1 | 1 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 1
Body temperature increased (Investigations) | 0 | 1 | 1
Atypical mycobacterium test positive (Investigations) | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Blood phosphorus abnormal (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 1
Forced expiratory volume increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Glucose tolerance test abnormal (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Pseudomonas test positive (Investigations) | 1 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 1
Sputum abnormal (Investigations) | 1 | 0 | 0
Urine calcium increased (Investigations) | 0 | 0 | 1
Vitamin E decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 1 | 0
Fatigue (General disorders) | 19 | 17 | 17
Pyrexia (General disorders) | 12 | 12 | 17
Asthenia (General disorders) | 3 | 5 | 3
Pain (General disorders) | 2 | 4 | 3
Chest discomfort (General disorders) | 1 | 3 | 3
Malaise (General disorders) | 1 | 2 | 3
Chills (General disorders) | 1 | 0 | 2
Drug intolerance (General disorders) | 0 | 0 | 3
Chest pain (General disorders) | 2 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 1
Drug interaction (General disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 0 | 1
Feeling abnormal (General disorders) | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 1
Implant site thrombosis (General disorders) | 0 | 0 | 1
Local swelling (General disorders) | 1 | 0 | 0
Medical device pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 25 | 28 | 29
Dizziness (Nervous system disorders) | 5 | 5 | 5
Sinus headache (Nervous system disorders) | 2 | 3 | 3
Migraine (Nervous system disorders) | 3 | 0 | 3
Lethargy (Nervous system disorders) | 1 | 2 | 2
Dysgeusia (Nervous system disorders) | 2 | 0 | 2
Poor quality sleep (Nervous system disorders) | 0 | 0 | 3
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 8 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 4
Acne (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Chloasma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Gout (Metabolism and nutrition disorders) | 2 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 3 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stoma site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 2 | 3
Anxiety (Psychiatric disorders) | 2 | 2 | 2
Depression (Psychiatric disorders) | 4 | 1 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 3
Irritability (Psychiatric disorders) | 1 | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Disturbance in social behaviour (Psychiatric disorders) | 0 | 0 | 1
Emotional disorder (Psychiatric disorders) | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0
Middle insomnia (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 1 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2 | 3
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 3
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 2 | 1
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Penile erythema (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 4 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 2 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 1 | 1
Ear canal erythema (Ear and labyrinth disorders) | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 2
Asthenopia (Eye disorders) | 1 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1 | 1
Astigmatism (Eye disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Eye disorder (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 0
Urine odour abnormal (Renal and urinary disorders) | 2 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 2
Flushing (Vascular disorders) | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Poor venous access (Vascular disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Defect conduction intraventricular (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 0 | 1
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.